CLINICAL TRIAL: NCT04126213
Title: A Phase II, Randomised, Observer-blind, Placebo Controlled Multi-country Study to Assess the Safety, Reactogenicity and Immunogenicity of a Single Intramuscular Dose of GSK Biologicals' Investigational RSV Maternal Unadjuvanted Vaccine (GSK3888550A), in Healthy Pregnant Women Aged 18 to 40 Years and Infants Born to Vaccinated Mothers
Brief Title: Study of Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline's (GSK)Respiratory Syncytial Virus (RSV)Maternal Unadjuvanted Vaccine in Healthy Pregnant Women (Aged 18 to 40 Years) and Their Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 209544; 2019-001991-12 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data was collected in an observer-blind manner. The laboratory in charge of the sample testing was blinded to the intervention assignment, codes were used to link the subject and study (without any link to the intervention attributed to the subject) to each sample. Investigators remained blinded to each subject's assigned study intervention until the second analysis. After the second analysis, the study was not considered observer blind as the investigator brochure was updated to include safety information presented by treatment group. This led to inadvertent unblinding of investigators and site staff to some subjects' treatment assignments. The subjects themselves remained blinded throughout their participation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- RSV MAT 60 Group-Mother (Experimental): Maternal subjects randomized to RSV MAT 60 Group received a single dose of RSV MAT (60 µg) vaccine at Day 1, and were followed up until the study end.
  Interventions: Biological: RSV MAT 60 µg
- RSV MAT 120 Group-Mother (Experimental): Maternal subjects randomized to RSV MAT 120 group received a single dose of RSV MAT (120 µg) vaccine at Day 1, and were followed up until the study end.
  Interventions: Biological: RSV MAT 120 µg
- Control Group-Mother (Placebo Comparator): Maternal subjects randomized to the Control Group received a single dose of Placebo at Day 1, and were followed up until the study end.
  Interventions: Drug: Placebo
- RSV MAT 60 Group-Infant (No Intervention): This group consisted of infants born to mothers (from RSV MAT 60 Group-Mother) who received a single dose of RSV MAT (60 µg) vaccine during pregnancy.
- RSV MAT 120 Group-Infant (No Intervention): This group consisted of infants born to mothers (from RSV MAT 120 Group-Mother) who received a single dose of RSV MAT (120 µg) vaccine during pregnancy.
- Control Group-Infant (No Intervention): This group consisted of infants born to mothers (from Control Group-Mother) who received a single dose of placebo during pregnancy.

INTERVENTIONS:
Biological: RSV MAT 60 µg — One single dose of RSV MAT 60 µg vaccine administered intramuscularly in the deltoid region of the non-dominant arm on Day 1.
  Arms: RSV MAT 60 Group-Mother
Biological: RSV MAT 120 µg — One single dose of RSV MAT 120 µg vaccine administered intramuscularly in the deltoid region of the non-dominant arm on Day 1.
  Arms: RSV MAT 120 Group-Mother
Drug: Placebo — One single dose of placebo (NaCl solution) administered intramuscularly in the deltoid region of the non-dominant arm on Day 1.
  Arms: Control Group-Mother

SUMMARY:
The purpose of this study was to evaluate the safety and immune response to a single intramuscular (IM) dose of GSK Biologicals' investigational RSV maternal vaccine (RSVPreF3) in healthy pregnant women 18-40 years of age and in infants born to vaccinated mothers.

ELIGIBILITY:
Inclusion Criteria:

Maternal subjects

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Subjects who give written or witnessed/thumb printed informed consent after the study has been explained according to local regulatory requirements, and before any study specific procedures are performed. The informed consent given at screening should (consistent with local regulations / guidelines) either:

  * include consent for both the maternal subject's participation and participation of the infant after the infant's birth, or
  * include consent for the maternal subject's participation and expressed willingness to consider permitting the infant to take part after the infant's birth.
  * Both mother and father should consent if local regulations/guidelines require it.
* Age 18 to 40 years, inclusive, when informed consent is given.
* Pre-pregnancy BMI 18.5 to 34.9, inclusive
* Healthy as established by medical history and clinical examination before entering into the study.
* At 28^0/7 to 33^6/7 weeks of gestation at the time of study vaccination (Visit 1), as established by last menstrual period (LMP) date corroborated by first or second trimester ultrasound examination (U/S).

  * If LMP and U/S do not correlate, default to U/S gestational age assessment. The level of diagnostic certainty of the gestational age should be established by using the Global Alignment of Immunisation safety Assessment in pregnancy gestation age assessment tool
* Subject satisfying screening requirements
* Singleton pregnancy
* HIV negative, as assessed by local standard of care serologic tests conducted during the current pregnancy and before enrolment (Visit 1).
* No fetal genetic abnormalities.
* No significant congenital malformations, as assessed by level 2 ultrasound (also known as a fetal anomaly ultrasound scan or fetal morphology assessment) conducted after 18 weeks of gestation
* Willing to provide cord blood
* Willing to have the infant followed-up after delivery for a period of 12 months
* Does not plan after delivery to give the infant for adoption or place the infant in care Note that women whose pregnancies resulted from Assisted Reproductive Technologies may be enrolled if they meet all inclusion criteria and none of the exclusion criteria.

Infant subjects

* Live-born from the study pregnancy.
* Re-signed (confirmed) written or witnessed/thumb printed informed consent for study participation of the infant obtained from the infant's mother and/or father and/or legally authorized representative, as applicable by local law, before performing any study specific procedure.

Exclusion Criteria:

Maternal subjects

Medical conditions

* History of allergic disease or reactions likely to be exacerbated by any component of the RSV vaccine
* Hypersensitivity to latex
* Significant complications in the current pregnancy such as:

  * Gestational hypertension at ≥20 weeks of gestation in the absence of proteinuria in a woman with a previously normal blood pressure
  * Gestational diabetes which is not controlled by diet and exercise
  * Pre-eclampsia
  * Eclampsia during current pregnancy
  * Intrauterine growth restriction
  * Placenta previa
  * Placental abruption, placenta accreta/percreta/increta, chorioamnionitis or any abnormalities that in the opinion of Investigator can impair the maternal-fetal circulation
  * Polyhydramnios
  * Oligohydramnios
  * Cervical suture in place
  * Preterm labour or history of preterm labour in the current pregnancy
  * Ongoing medical intervention to prevent preterm delivery or medical treatment for suspected preterm delivery
  * Cholestasis
  * Other pregnancy-related complications that in the Investigator's judgement would preclude participation of the subjects in an investigational vaccine trial or might pose risk to the subject due to participation in the study
* Significant structural abnormalities of the uterus or cervix
* History of prior stillbirth or neonatal death
* History of preterm birth
* History of ≥2 spontaneous abortions
* Known or suspected HBV or HCV infection, based on medical history and clinical presentation
* Known or suspected infection during the current pregnancy with Toxoplasma, Parvovirus B19, Syphilis, Zika, Rubella, Varicella, CMV or primary genital Herpes Simplex, based on medical history and clinical presentation
* Active infection with tuberculosis, based on medical history and clinical presentation
* Known or suspected impairment of the immune system or autoimmune disorder (based on medical history and physical examination; no laboratory testing required)
* Lymphoproliferative disorder or malignancy within 5 years before vaccination (excluding effectively treated non-melanoma skin cancer)
* Any clinically significant grade 1 hematological and/or biochemical laboratory abnormalities identified at screening, which are clinically significant for pregnant women in the second and third trimester
* Grade ≥ 2 hematological and/or biochemical laboratory abnormalities identified at screening being clinically significant for pregnant women in the second and third trimester
* Acute or chronic clinically significant conditions, that might pose additional risk to the subject due to participation in the study
* Any conditions that, may interfere with subject's ability to comply with study procedures or receipt of prenatal care
* Any condition which, would increase the risks of study participation to the unborn infant

Prior/Concomitant therapy

* Prior receipt of a COVID-19 vaccine.
* Prior receipt of an RSV vaccine
* Use of any investigational or non-registered product other than the study vaccine(s)/product(s) during the period beginning 29 days before the dose of study vaccine/product or planned use during the study period
* Planned administration/administration of any vaccine within 29 days before study vaccine administration and through Day 43 post-delivery, except seasonal influenza vaccines and dTpa/Tdap or tetanus, which may be administered according to standard of care ≥ 15 days before or after study vaccination
* Administration of immunoglobulins, blood products or plasma derivatives within 3 months before study vaccination or planned administration through Visit 5
* Administration of immune-modifying therapy within 6 months before the study vaccine/product dose, or planned administration through delivery. This includes but is not limited to:

  * Azathioprine, mycophenolate mofetil, 6-mercaptopurine, cyclosporine, tacrolimus, monoclonal or polyclonal antibodies;
  * Prednisone, ≥ 5 mg/day or equivalent for ≥ 14 days. Topical, steroids are allowed. Inhaled steroids are allowed if ≤ 500µg/day of beclomethasone or fluticasone, or ≤ 800µg/day of budesonide.

Prior/Concomitant clinical study experience

* Previous participation in a clinical trial of an RSV vaccine
* Concurrently participating in another clinical study, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product

Other exclusions

* Alcoholism or substance use disorder within the past 24 months based on the presence of two or more abuse criteria
* A local condition that precludes injection of the study drug or precludes assessment of local reactogenicity
* Consanguinity of maternal subject and her partner (second degree cousins or closer)
* Any study personnel or their immediate dependants, family, or household members

Infant subjects

* Concurrently participating in another clinical study, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Child in care

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 534 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (13):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Englewood, Ohio
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Plano, Texas
- Australia (2):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Melbourne, Victoria
- Canada (2):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Québec
- GSK Investigational Site, Helsinki, Finland
- France (2):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Saint-Etienne
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Soweto, Gauteng, South Africa
- Spain (6):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Marbella

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bebia Z, Reyes O, Jeanfreau R, Kantele A, De Leon RG, Sanchez MG, Banooni P, Gardener GJ, Rasero JLB, Pardilla MBE, Langley JM, Di Leo CM, Botelho-Nevers E, Buttery J, Laurichesse H, Madhi SA, Garcia AM, Stanley T, Barjat T, Griffith R, Castrejon-Alba MM, de Heusch M, Dieussaert I, Hercor M, Lese P, Qian H, Tullio AN, Henry O. Safety and Immunogenicity of an Investigational Respiratory Syncytial Virus Vaccine (RSVPreF3) in Mothers and Their Infants: A Phase 2 Randomized Trial. J Infect Dis. 2023 Aug 11;228(3):299-310. doi: 10.1093/infdis/jiad024. PMID 36722147

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 534 participants who signed the informed consent 213 maternal subjects were vaccinated, and 206 infants were born to those exposed mothers. Therefore, a total of 419 are considered exposed.
Period: Overall Study
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Started | 70 | 75 | 68 | 67 | 73 | 66
Completed | 58 | 70 | 59 | 54 | 67 | 55
Not Completed | 12 | 5 | 9 | 13 | 6 | 11
Not completed — Lost to Follow-up | 9 | 1 | 5 | 10 | 4 | 7
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 2 | 2 | 0 | 1
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 2 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant | Total
Number analyzed (Participants) | 70 | 75 | 68 | 67 | 73 | 66 | 419
Age, Customized [Count of Participants; unit: Participants]
  0 to 1 years | 0 | 0 | 0 | 67 | 73 | 66 | 206
  18 < 35 years | 59 | 62 | 56 | 0 | 0 | 0 | 177
  >= 35 years | 11 | 13 | 12 | 0 | 0 | 0 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 75 | 68 | 28 | 30 | 37 | 308
  Male | 0 | 0 | 0 | 39 | 43 | 29 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 2 | 0 | 0 | 1 | 0 | 3
  ASIAN | 0 | 0 | 2 | 0 | 0 | 1 | 3
  BLACK OR AFRICAN AMERICAN | 12 | 12 | 13 | 12 | 9 | 9 | 67
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 3 | 1 | 0 | 3 | 2 | 1 | 10
  OTHER | 10 | 10 | 7 | 10 | 11 | 8 | 56
  UNKNOWN | 0 | 2 | 1 | 0 | 1 | 1 | 5
  WHITE | 45 | 48 | 45 | 42 | 49 | 46 | 275

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Maternal Subjects With Any Solicited Administration Site Events
Description: Assessed solicited administration site events were pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Any erythema and swelling symptom = symptom reported with a surface diameter greater than 0 millimeters.
Time Frame: During the 7-day follow-up period after vaccination (i.e. day of vaccination and 6 subsequent days)
Population: The analysis was performed on the Solicited Safety Set (SSS), which included all the maternal subjects who received at least 1 dose of the study intervention and who had solicited safety data.
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 66
Percentage of maternal subjects
  Any Pain | 57.1 [44.7 to 68.9] | 52 [40.2 to 63.7] | 15.2 [7.5 to 26.1]
  Any Erythema | 1.4 [0 to 7.7] | 6.7 [2.2 to 14.9] | 0 [0 to 5.4]
  Any Swelling | 4.3 [0.9 to 12] | 4 [0.8 to 11.2] | 0 [0 to 5.4]

2. Primary Outcome: Percentage of Maternal Subjects With Any Solicited Systemic Events
Description: Assessed solicited systemic events were fatigue, headache, nausea, vomiting, diarrhea, abdominal pain and fever [temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relation to study intervention.
Time Frame: During the 7-day follow-up period after vaccination (i.e. day of vaccination and 6 subsequent days)
Population: The analysis was performed on the SSS, which included all the maternal subjects who received at least 1 dose of the study intervention and who had solicited safety data.
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 66
Percentage of maternal subjects
  Any Fatigue | 40 [28.5 to 52.4] | 34.7 [24 to 46.5] | 25.8 [15.8 to 38]
  Any Headache | 34.3 [23.3 to 46.6] | 28 [18.2 to 39.6] | 19.7 [10.9 to 31.3]
  Any Nausea | 25.7 [16 to 37.6] | 22.7 [13.8 to 33.8] | 13.6 [6.4 to 24.3]
  Any Vomiting | 7.1 [2.4 to 15.9] | 9.3 [3.8 to 18.3] | 4.5 [0.9 to 12.7]
  Any Diarrhea | 14.3 [7.1 to 24.7] | 17.3 [9.6 to 27.8] | 13.6 [6.4 to 24.3]
  Any Abdominal pain | 12.9 [6.1 to 23] | 22.7 [13.8 to 33.8] | 9.1 [3.4 to 18.7]
  Any Fever | 0 [0 to 5.1] | 0 [0 to 4.8] | 0 [0 to 5.4]

3. Primary Outcome: Number of Maternal Subjects With Any Haematological Laboratory Abnormalities at Day 8 by Baseline Ranges
Description: Hematological parameters assessed were Eosinophils (EOS), Erythrocytes (ERY), Hematocrit (HEM), Lymphocytes (LYMP), Mean Corpuscular Volume (MCV), Neutrophils (NEU), Platelets (PLA), and White Blood Cells (WBC) count. The increase and/or decrease of these parameters were evaluated at Day 8. Abnormal laboratory values refer to range indicator at Day 8 (D8) categorized as Missing, Below, Within and Above normal values and compared to the baseline (B) range indicator of the same parameter, at Screening (up to 15 days before vaccination) i.e. Missing, Below, Within and Above. E.g. 'WBC decrease Below (B) - Within (D8)' = WBC decrease in subjects with below normal values at baseline and within normal values at Day 8.
Time Frame: At Day 8
Population: The analysis was performed on the Exposed Set-Maternal (ESM), which included all the maternal subjects who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Participants
  EOS Increase Below (B)-Below (D8) | 6 | 5 | 2
  EOS Increase Below (B)-Within (D8) | 6 | 2 | 4
  EOS Increase Below (B)-Above (D8) | 0 | 0 | 0
  EOS Increase Below (B)-Unknown (D8) | 0 | 0 | 1
  EOS Increase Within (B)-Below (D8) | 2 | 5 | 2
  EOS Increase Within (B)-Within (D8) | 53 | 58 | 56
  EOS Increase Within (B)-Above (D8) | 0 | 0 | 0
  EOS Increase Within (B)-Unknown (D8) | 2 | 3 | 1
  EOS Increase Above (B)-Below (D8) | 0 | 0 | 0
  EOS Increase Above (B)-Within (D8) | 0 | 1 | 0
  EOS Increase Above (B)-Above (D8) | 1 | 1 | 0
  EOS Increase Above (B)-Unknown (D8) | 0 | 0 | 0
  EOS Increase Unknown(B)-Below (D8) | 0 | 0 | 0
  EOS Increase Unknown (B)-Within (D8) | 0 | 0 | 2
  EOS Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  EOS Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  ERY Decrease Below (B)-Below (D8) | 24 | 35 | 23
  ERY Decrease Below (B)-Within (D8) | 4 | 2 | 5
  ERY Decrease Below (B)-Above (D8) | 0 | 0 | 0
  ERY Decrease Below (B)-Unknown (D8) | 1 | 2 | 2
  ERY Decrease Within (B)-Below (D8) | 6 | 2 | 7
  ERY Decrease Within (B)-Within (D8) | 34 | 34 | 29
  ERY Decrease Within (B)-Above (D8) | 0 | 0 | 0
  ERY Decrease Within(B)-Unknown (D8) | 1 | 0 | 0
  ERY Decrease Above (B)-Below (D8) | 0 | 0 | 0
  ERY Decrease Above (B)-Within (D8) | 0 | 0 | 0
  ERY Decrease Above (B)-Above (D8) | 0 | 0 | 0
  ERY Decrease Above (B)-Unknown (D8) | 0 | 0 | 0
  ERY Decrease Unknown (B)-Below (D8) | 0 | 0 | 2
  ERY Decrease Unknown (B)-Within (D8) | 0 | 0 | 0
  ERY Decrease Unknown (B)-Above (D8) | 0 | 0 | 0
  ERY Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  ERY Increase Below (B)-Below (D8) | 24 | 35 | 23
  ERY Increase Below (B)-Within (D8) | 4 | 2 | 5
  ERY Increase Below (B)-Above (D8) | 0 | 0 | 0
  ERY Increase Below (B)-Unknown (D8) | 1 | 2 | 2
  ERY Increase Within (B)-Below (D8) | 6 | 2 | 7
  ERY Increase Within (B)-Within (D8) | 34 | 34 | 29
  ERY Increase Within (B)-Above (D8) | 0 | 0 | 0
  ERY Increase Within (B)-Unknown (D8) | 1 | 0 | 0
  ERY Increase Above-Below (D8) | 0 | 0 | 0
  ERY Increase Above (B)-Within (D8) | 0 | 0 | 0
  ERY Increase Above (B)-Above (D8) | 0 | 0 | 0
  ERY Increase Above (B)-Unknown (D8) | 0 | 0 | 0
  ERY Increase Unknown (B)-Below (D8) | 0 | 0 | 2
  ERY Increase Unknown (B)-Within (D8) | 0 | 0 | 0
  ERY Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  ERY Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  HEM Decrease Below (B)-Below (D8) | 25 | 26 | 24
  HEM Decrease Below (B)-Within (D8) | 2 | 3 | 2
  HEM Decrease Below (B)-Above (D8) | 0 | 0 | 0
  HEM Decrease Below (B)-Unknown (D8) | 1 | 1 | 1
  HEM Decrease Within (B)-Below (D8) | 7 | 9 | 7
  HEM Decrease Within (B)- Within (D8) | 34 | 35 | 31
  HEM Decrease Within (B)-Above (D8) | 0 | 0 | 0
  HEM Decrease Within (B)-Unknown (D8) | 1 | 1 | 1
  HEM Decrease Above (B)-Below (D8) | 0 | 0 | 0
  HEM Decrease Above (B)-Within (D8) | 0 | 0 | 0
  HEM Decrease Above (B)-Above (D8) | 0 | 0 | 0
  HEM Decrease Above (B)-Unknown (D8) | 0 | 0 | 0
  HEM Decrease Unknown (B)-Below (D8) | 0 | 0 | 2
  HEM Decrease Unknown (B)-Within (D8) | 0 | 0 | 0
  HEM Decrease Unknown (B)-Above (D8) | 0 | 0 | 0
  HEM Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  HEM Increase Below (B)-Below (D8) | 25 | 26 | 24
  HEM Increase Below (B)-Within (D8) | 2 | 3 | 2
  HEM Increase Below (B)-Above (D8) | 0 | 0 | 0
  HEM Increase Below (B)-Unknown (D8) | 1 | 1 | 1
  HEM Increase Within (B)-Below (D8) | 7 | 9 | 7
  HEM Increase Within (B)-Within (D8) | 34 | 35 | 31
  HEM Increase Within (B)-Above (D8) | 0 | 0 | 0
  HEM Increase Within (B)-Unknown (D8) | 1 | 1 | 1
  HEM Increase Above (B)-Below (D8) | 0 | 0 | 0
  HEM Increase Above (B)-Within (D8) | 0 | 0 | 0
  HEM Increase Above (B)-Above (D8) | 0 | 0 | 0
  HEM Increase Above (B)-Unknown (D8) | 0 | 0 | 0
  HEM Increase Unknown (B)-Below (D8) | 0 | 0 | 2
  HEM Increase Unknown (B)-Within (D8) | 0 | 0 | 0
  HEM Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  HEM Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Decrease Below (B)-Below (D8) | 0 | 0 | 0
  LYMP Decrease Below (B)-Within (D8) | 0 | 0 | 1
  LYMP Decrease Below (B)-Above (D8) | 0 | 0 | 0
  LYMP Decrease Below (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Decrease Within (B)-Below (D8) | 0 | 0 | 0
  LYMP Decrease Within (B)-Within (D8) | 68 | 72 | 63
  LYMP Decrease Within (B)-Above (D8) | 0 | 0 | 0
  LYMP Decrease Within (B)-Unknown (D8) | 2 | 3 | 2
  LYMP Decrease Above (B)-Below (D8) | 0 | 0 | 0
  LYMP Decrease Above (B)-Within (D8) | 0 | 0 | 0
  LYMP Decrease Above (B)-Above (D8) | 0 | 0 | 0
  LYMP Decrease Above (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Decrease Unknown (B)-Below (D8) | 0 | 0 | 0
  LYMP Decrease Unknown (B)-Within (D8) | 0 | 0 | 2
  LYMP Decrease Unknown (B)-Above (D8) | 0 | 0 | 0
  LYMP Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Increase Below (B)-Below (D8) | 0 | 0 | 0
  LYMP Increase Below (B)-Within (D8) | 0 | 0 | 1
  LYMP Increase Below (B)-Above (D8) | 0 | 0 | 0
  LYMP Increase Below (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Increase Within (B)-Below (D8) | 0 | 0 | 0
  LYMP Increase Within (B)-Within (D8) | 68 | 72 | 63
  LYMP Increase Within (B)-Above (D8) | 0 | 0 | 0
  LYMP Increase Within (B)-Unknown (D8) | 2 | 3 | 2
  LYMP Increase Above (B)-Below (D8) | 0 | 0 | 0
  LYMP Increase Above (B)-Within (D8) | 0 | 0 | 0
  LYMP Increase Above (B)-Above (D8) | 0 | 0 | 0
  LYMP Increase Above (B)-Unknown (D8) | 0 | 0 | 0
  LYMP Increase Unknown (B)-Below (D8) | 0 | 0 | 0
  LYMP Increase Unknown (B)-Within (D8) | 0 | 0 | 2
  LYMP Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  LYMP Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  MCV Decrease Below (B)-Below (D8) | 2 | 1 | 1
  MCV Decrease Below (B)-Within (D8) | 0 | 0 | 0
  MCV Decrease Below (B)-Above (D8) | 0 | 0 | 0
  MCV Decrease Below (B)-Unknown (D8) | 0 | 0 | 0
  MCV Decrease Within (B)-Below (D8) | 0 | 0 | 1
  MCV Decrease Within (B)-Within (D8) | 62 | 66 | 57
  MCV Decrease Within (B)-Above (D8) | 2 | 2 | 1
  MCV Decrease Within (B)-Unknown (D8) | 2 | 1 | 2
  MCV Decrease Above (B)-Below (D8) | 0 | 0 | 0
  MCV Decrease Above (B)-Within (D8) | 0 | 2 | 1
  MCV Decrease Above (B)-Above (D8) | 2 | 2 | 3
  MCV Decrease Above (B)-Unknown (D8) | 0 | 1 | 0
  MCV Decrease Unknown (B)-Below (D8) | 0 | 0 | 0
  MCV Decrease Unknown (B)-Within (D8) | 0 | 0 | 2
  MCV Decrease Unknown (B)-Above (D8) | 0 | 0 | 0
  MCV Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  MCV Increase Below (B)-Below (D8) | 2 | 1 | 1
  MCV Increase Below (B)-Within (D8) | 0 | 0 | 0
  MCV Increase Below (B)-Above (D8) | 0 | 0 | 0
  MCV Increase Below (B)- Unknown (D8) | 0 | 0 | 0
  MCV Increase Within (B)-Below (D8) | 0 | 0 | 1
  MCV Increase Within (B)-Within (D8) | 62 | 66 | 57
  MCV Increase Within (B)-Above (D8) | 2 | 2 | 1
  MCV Increase Within (B)-Unknown (D8) | 2 | 1 | 2
  MCV Increase Above (B)-Below (D8) | 0 | 0 | 0
  MCV Increase Above (B)-Within (D8) | 0 | 2 | 1
  MCV Increase Above (B)-Above (D8) | 2 | 2 | 3
  MCV Increase Above (B)-Unknown (D8) | 0 | 1 | 0
  MCV Increase Unknown (B)-Below (D8) | 0 | 0 | 0
  MCV Increase Unknown (B)-Within (D8) | 0 | 0 | 2
  MCV Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  MCV Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  NEU Decrease Below (B)-Below (D8) | 0 | 0 | 0
  NEU Decrease Below (B)-Within (D8) | 0 | 0 | 0
  NEU Decrease Below (B)-Above (D8) | 0 | 0 | 0
  NEU Decrease Below (B)-Unknown (D8) | 0 | 0 | 0
  NEU Decrease Within (B)-Below (D8) | 0 | 0 | 0
  NEU Decrease Within (B)-Within (D8) | 42 | 46 | 41
  NEU Decrease Within (B)-Above (D8) | 8 | 9 | 9
  NEU Decrease Within (B)-Unknown (D8) | 0 | 2 | 1
  NEU Decrease Above (B)-Below (D8) | 0 | 0 | 0
  NEU Decrease Above (B)-Within (D8) | 5 | 5 | 6
  NEU Decrease Above (B)-Above (D8) | 13 | 12 | 8
  NEU Decrease Above (B)-Unknown (D8) | 2 | 1 | 1
  NEU Decrease Unknown (B)-Below (D8) | 0 | 0 | 0
  NEU Decrease Unknown (B)-Within (D8) | 0 | 0 | 1
  NEU Decrease Unknown (B)-Above (D8) | 0 | 0 | 1
  NEU Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  PLA Decrease Below (B)-Below (D8) | 0 | 0 | 0
  PLA Decrease Below (B)-Within (D8) | 1 | 1 | 0
  PLA Decrease Below (B)-Above (D8) | 0 | 0 | 0
  PLA Decrease Below (B)-Unknown (D8) | 0 | 0 | 0
  PLA Decrease Within (B)-Below (D8) | 0 | 0 | 0
  PLA Decrease Within (B)-Within (D8) | 67 | 72 | 63
  PLA Decrease Within (B)-Above (D8) | 0 | 0 | 0
  PLA Decrease Within (B)-Unknown (D8) | 2 | 2 | 2
  PLA Decrease Above (B)-Below (D8) | 0 | 0 | 0
  PLA Decrease Above (B)-Within (D8) | 0 | 0 | 1
  PLA Decrease Above (B)- Above (D8) | 0 | 0 | 0
  PLA Decrease Above (B)-Unknown (D8) | 0 | 0 | 0
  PLA Decrease Unknown (B)-Below (D8) | 0 | 0 | 0
  PLA Decrease Unknown (B)-Within (D8) | 0 | 0 | 2
  PLA Decrease Unknown (B)-Above (D8) | 0 | 0 | 0
  PLA Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  PLA Increase Below (B)-Below (D8) | 0 | 0 | 0
  PLA Increase Below (B)-Within (D8) | 1 | 1 | 0
  PLA Increase Below (B)-Above (D8) | 0 | 0 | 0
  PLA Increase, Below (B)-Unknown (D8) | 0 | 0 | 0
  PLA Increase Within (B)-Below (D8) | 0 | 0 | 0
  PLA Increase Within (B)-Within (D8) | 67 | 72 | 63
  PLA Increase Within (B)-Above (D8) | 0 | 0 | 0
  PLA Increase Within (B)-Unknown (D8) | 2 | 2 | 2
  PLA Increase Above (B)-Below (D8) | 0 | 0 | 0
  PLA Increase Above (B)-Within (D8) | 0 | 0 | 1
  PLA Increase Above (B)-Above (D8) | 0 | 0 | 0
  PLA Increase Above (B)-Unknown (D8) | 0 | 0 | 0
  PLA Increase Unknown (B)-Below (D8) | 0 | 0 | 0
  PLA Increase Unknown (B)-Within (D8) | 0 | 0 | 2
  PLA Increase Unknown (B)-Above (D8) | 0 | 0 | 0
  PLA Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  WBC Decrease Below (B)-Below (D8) | 0 | 0 | 0
  WBC Decrease Below (B)-Within (D8) | 0 | 0 | 0
  WBC Decrease Below (B)-Above (D8) | 0 | 0 | 0
  WBC Decrease Below (B)-Unknown (D8) | 0 | 0 | 0
  WBC Decrease Within (B)-Below (D8) | 0 | 0 | 0
  WBC Decrease Within (B)-Within (D8) | 46 | 48 | 46
  WBC Decrease Within (B)-Above (D8) | 5 | 8 | 5
  WBC Decrease Within (B)-Unknown (D8) | 1 | 1 | 2
  WBC Decrease Above (B)-Below (D8) | 0 | 0 | 0
  WBC Decrease Above (B)-Within (D8) | 3 | 5 | 3
  WBC Decrease Above (B)-Above (D8) | 14 | 12 | 10
  WBC Decrease Above (B)-Unknown (D8) | 1 | 1 | 0
  WBC Decrease Unknown (B)-Below (D8) | 0 | 0 | 0
  WBC Decrease Unknown (B)-Within (D8) | 0 | 0 | 1
  WBC Decrease Unknown (B)-Above (D8) | 0 | 0 | 1
  WBC Decrease Unknown (B)-Unknown (D8) | 0 | 0 | 0
  WBC Increase Below (B)-Below (D8) | 0 | 0 | 0
  WBC Increase Below (B)-Within (D8) | 0 | 0 | 0
  WBC Increase Below (B)-Above (D8) | 0 | 0 | 0
  WBC Increase Below (B)-Unknown (D8) | 0 | 0 | 0
  WBC Increase Within (B)-Below (D8) | 0 | 0 | 0
  WBC Increase Within (B)-Within (D8) | 46 | 48 | 46
  WBC Increase Within (B)- Above (D8) | 5 | 8 | 5
  WBC Increase Within (B)-Unknown (D8) | 1 | 1 | 2
  WBC Increase Above (B)-Below (D8) | 0 | 0 | 0
  WBC Increase Above (B)-Within (D8) | 3 | 5 | 3
  WBC Increase Above (B)-Above (D8) | 14 | 12 | 10
  WBC Increase Above (B)- Unknown (D8) | 1 | 1 | 0
  WBC Increase Unknown (B)-Below (D8) | 0 | 0 | 0
  WBC Increase Unknown (B)-Within (D8) | 0 | 0 | 1
  WBC Increase Unknown (B)-Above (D8) | 0 | 0 | 1
  WBC Increase Unknown (B)-Unknown (D8) | 0 | 0 | 0

4. Primary Outcome: Number of Maternal Subjects With Any Biochemical Laboratory Abnormalities at Day 8 by Baseline Ranges
Description: Biochemical parameters assessed were Alanine Amino-Transferase (ALT), Aspartate Amino-Transferase (AST), Creatinine (CRE) and Urea nitrogen (URN). The increase was evaluated only for AST and ALT parameters at Day 8. Abnormal laboratory values refer to range indicator at Day 8 (D8) categorized as Missing, Below, Within and Above normal values and compared to the baseline (B) range indicator of the same parameter, at Screening (up to 15 days before vaccination) i.e. Missing, Below, Within and Above. E.g. 'AST increase Below (B) - Within (D8)' = AST increase in subjects with below normal values at baseline and within normal values at Day 8.
Time Frame: At Day 8
Population: The analysis was performed on the ESM, which included all the maternal subjects who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Participants
  ALT increase Below (B)-Below (D8) | 0 | 0 | 0
  ALT increase Below (B)- Within (D8) | 0 | 0 | 0
  ALT increase Below (B)- Above (D8) | 0 | 0 | 0
  ALT increase Below (B)-Unknown (D8) | 0 | 0 | 0
  ALT increase Within (B)- Below (D8) | 0 | 0 | 0
  ALT increase Within (B)-Within (D8) | 64 | 69 | 65
  ALT increase Within (B)- Above (D8) | 1 | 0 | 0
  ALT increase Within (B)-Unknown (D8) | 2 | 3 | 1
  ALT increase Above (B)- Below (D8) | 0 | 0 | 0
  ALT increase Above (B)- Within (D8) | 1 | 2 | 0
  ALT increase Above (B)- Above (D8) | 1 | 1 | 0
  ALT increase Above (B)-Unknown (D8) | 0 | 0 | 0
  ALT increase Unknown (B)-Below (D8) | 0 | 0 | 0
  ALT increase Unknown (B)-Within (D8) | 1 | 0 | 2
  ALT increase Unknown (B)-Above (D8) | 0 | 0 | 0
  ALT increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  AST increase Below (B)-Below (D8) | 0 | 0 | 0
  AST increase Below (B)- Within (D8) | 0 | 0 | 0
  AST increase Below (B)- Above (D8) | 0 | 0 | 0
  AST increase Below (B)-Unknown (D8) | 0 | 0 | 0
  AST increase Within (B)- Below (D8) | 0 | 0 | 0
  AST increase Within (B)-Within (D8) | 67 | 71 | 65
  AST increase Within (B)- Above (D8) | 0 | 1 | 0
  AST increase Within (B)-Unknown (D8) | 1 | 2 | 1
  AST increase Above (B)- Below (D8) | 0 | 0 | 0
  AST increase Above (B)-Within (D8) | 0 | 1 | 0
  AST increase Above (B)-Above (D8) | 1 | 0 | 0
  AST increase Above (B)-Unknown (D8) | 0 | 0 | 0
  AST increase Unknown (B)-Below (D8) | 0 | 0 | 0
  AST increase Unknown (B)-Within (D8) | 1 | 0 | 2
  AST increase Unknown (B)-Above (D8) | 0 | 0 | 0
  AST increase Unknown (B)-Unknown (D8) | 0 | 0 | 0
  Creatinine Below (B)-Below (D8) | 16 | 18 | 18
  Creatinine Below (B)-Within (D8) | 6 | 9 | 4
  Creatinine Below (B)-Above (D8) | 0 | 0 | 0
  Creatinine Below (B)- Unknown (D8) | 0 | 0 | 1
  Creatinine Within (B)-Below (D8) | 2 | 4 | 6
  Creatinine Within (B)-Within (D8) | 45 | 42 | 37
  Creatinine Within (B)-Above (D8) | 0 | 0 | 0
  Creatinine Within (B)-Unknown (D8) | 1 | 2 | 0
  Creatinine Above (B)-Below (D8) | 0 | 0 | 0
  Creatinine Above (B)-Within (D8) | 0 | 0 | 0
  Creatinine Above (B)-Above (D8) | 0 | 0 | 0
  Creatinine Above (B)-Unknown (D8) | 0 | 0 | 0
  Creatinine Unknown (B)-Below (D8) | 0 | 0 | 1
  Creatinine Unknown (B)-Within (D8) | 0 | 0 | 1
  Creatinine Unknown (B)-Above (D8) | 0 | 0 | 0
  Creatinine Unknown (B)-Unknown (D8) | 0 | 0 | 0
  URN Below (B)-Below (D8) | 13 | 15 | 13
  URN Below (B)-Within (D8) | 6 | 4 | 3
  URN Below (B)-Above (D8) | 0 | 0 | 0
  URN Below (B)-Unknown (D8) | 0 | 1 | 1
  URN Within (B)-Below (D8) | 5 | 4 | 9
  URN Within (B)-Within (D8) | 45 | 49 | 39
  URN Within (B)-Above (D8) | 0 | 0 | 0
  URN Within (B)-Unknown (D8) | 1 | 1 | 0
  URN Above (B)-Below (D8) | 0 | 0 | 0
  URN Above (B)-Within (D8) | 0 | 0 | 0
  URN Above (B)-Above (D8) | 0 | 0 | 0
  URN Above (B)-Unknown (D8) | 0 | 0 | 0
  URN Unknown (B)-Below (D8) | 0 | 0 | 0
  URN Unknown (B)-Within (D8) | 0 | 1 | 3
  URN Unknown (B)-Above (D8) | 0 | 0 | 0
  URN Unknown (B)-Unknown (D8) | 0 | 0 | 0

5. Primary Outcome: Percentage of Maternal Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AE is any AE reported in addition to those solicited during the clinical study and that was spontaneously communicated by a maternal subject. Also, any solicited symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited AE. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days)
Population: The analysis was performed on the Unsolicited Safety Set-Maternal, which included maternal subjects who received at least 1 dose of the study intervention (ESM) that reported unsolicited AEs/reported not having unsolicited AEs.
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 30 [19.6 to 42.1] | 33.3 [22.9 to 45.2] | 33.8 [22.8 to 46.3]

6. Primary Outcome: Percentage of Maternal Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed included any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study subject or abnormal pregnancy outcomes (spontaneous abortion, foetal death, stillbirth, congenital anomalies, ectopic pregnancy), other situations (medical events that might jeopardize the participant or required medical/surgical intervention to prevent one of the other SAEs listed above: e.g. invasive/malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization). Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From Day 1 to Day 43 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 22.9 [13.7 to 34.4] | 26.7 [17.1 to 38.1] | 22.1 [12.9 to 33.8]

7. Primary Outcome: Percentage of Maternal Subjects With AEs Leading to Study Withdrawal
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs leading to study withdrawal = AEs identified by investigators to cause subject(s) withdrawal until the resolution of the event. These subject withdrawals were considered different from subject withdrawals for other reasons.
Time Frame: From Day 1 to Day 43 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

8. Primary Outcome: Percentage of Maternal Subjects With Any Medically Attended AEs (MAE)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Also, for instances where, due to the special circumstances, the subject could not seek medical advice for symptoms/an illness by visiting a medical facility or arranging for a home visit, the subject sought this advice instead via telephone, SMS, email, videotelephony or telemedicine, or other means. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From Day 1 to Day 43 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 41.4 [29.8 to 53.8] | 48 [36.3 to 59.8] | 42.6 [30.7 to 55.2]

9. Primary Outcome: Percentage of Maternal Subjects With Pregnancy Outcomes
Description: Pregnancy outcomes were: live birth with no congenital anomalies, live birth with congenital anomalies, Fetal death/still birth with no Congenital Anomalies (CA) - Antepartum and Unknown (Subjects withdrew from the study before delivery and pregnancy outcome information was not available for them).
Time Frame: From Day 1 to Day 43 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects
  Live birth with no congenital anomalies | 84.3 [73.6 to 91.9] | 81.3 [70.7 to 89.4] | 80.9 [69.5 to 89.4]
  Live birth with congenital anomalies | 12.9 [6.1 to 23] | 16 [8.6 to 26.3] | 16.2 [8.4 to 27.1]
  Fetal death/still birth with no CA- Antepartum | 0 [0 to 5.1] | 0 [0 to 4.8] | 1.5 [0 to 7.9]
  Unknown | 2.9 [0.3 to 9.9] | 2.7 [0.3 to 9.3] | 1.5 [0 to 7.9]

10. Primary Outcome: Percentage of Maternal Subjects With Pregnancy-related Adverse Events of Special Interest (AESIs)
Description: Pregnancy-related AESIs were: Non-Reassuring Fetal Status, Hypertensive Disorders of Pregnancy (HDP), Oligohydramnios, Pathways to Preterm Birth (PPB), Chorioamnionitis, Fetal Growth Restriction, Gestational Liver Disease (GLD), Postpartum Haemorrhage and Gestational Diabetes Mellitus.
Time Frame: From Day 1 to Day 43 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects
  Non-Reassuring Fetal Status | 8.6 [3.2 to 17.7] | 12 [5.6 to 21.6] | 11.8 [5.2 to 21.9]
  HDP-Gestational Hypertension | 4.3 [0.9 to 12] | 2.7 [0.3 to 9.3] | 1.5 [0 to 7.9]
  HDP-Pre-Eclampsia | 5.7 [1.6 to 14] | 2.7 [0.3 to 9.3] | 0 [0 to 5.3]
  Oligohydramnios | 4.3 [0.9 to 12] | 2.7 [0.3 to 9.3] | 1.5 [0 to 7.9]
  PPB-Preterm Labor | 0 [0 to 5.1] | 2.7 [0.3 to 9.3] | 2.9 [0.4 to 10.2]
  PPB-Preterm Rupture Of Membranes | 1.4 [0 to 7.7] | 0 [0 to 4.8] | 1.5 [0 to 7.9]
  PPB-Provider-Initiated Preterm Birth | 0 [0 to 5.1] | 1.3 [0 to 7.2] | 0 [0 to 5.3]
  Chorioamnionitis | 2.9 [0.3 to 9.9] | 2.7 [0.3 to 9.3] | 1.5 [0 to 7.9]
  Fetal Growth Restriction | 1.4 [0 to 7.7] | 2.7 [0.3 to 9.3] | 0 [0 to 5.3]
  GLD-Intrahepatic Cholestasis Of Pregnancy | 2.9 [0.3 to 9.9] | 1.3 [0 to 7.2] | 0 [0 to 5.3]
  Postpartum Haemorrhage | 1.4 [0 to 7.7] | 0 [0 to 4.8] | 1.5 [0 to 7.9]
  Gestational Diabetes Mellitus | 1.4 [0 to 7.7] | 0 [0 to 4.8] | 0 [0 to 5.3]

11. Primary Outcome: Percentage of Infant Subjects With Neonatal AESIs
Description: Neonatal AESIs, reported up to 6 weeks after birth were: Respiratory Distress In The Neonate, Macrosomia, Low Birth Weight, Small For Gestational Age, Preterm Birth, Large For Gestational Age, Neonatal Invasive Blood Stream Infections (NIBSI) and Congenital Anomalies (CA).
Time Frame: From birth to Day 43 post-birth
Population: The analysis was performed on the Exposed Set-Infant (ESI), which included all the infants live-born to exposed maternal subjects, whose parents/LARs completed the informed consent process and signed the informed consent form.
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects
  Respiratory Distress In The Neonate | 6 [1.7 to 14.6] | 6.8 [2.3 to 15.3] | 6.1 [1.7 to 14.8]
  Macrosomia | 3 [0.4 to 10.4] | 2.7 [0.3 to 9.5] | 7.6 [2.5 to 16.8]
  Low Birth Weight | 1.5 [0 to 8] | 5.5 [1.5 to 13.4] | 3 [0.4 to 10.5]
  Small For Gestational Age | 3 [0.4 to 10.4] | 4.1 [0.9 to 11.5] | 3 [0.4 to 10.5]
  Preterm Birth | 1.5 [0 to 8] | 4.1 [0.9 to 11.5] | 3 [0.4 to 10.5]
  Large For Gestational Age | 3 [0.4 to 10.4] | 0 [0 to 4.9] | 4.5 [0.9 to 12.7]
  NIBSI: Bacterial/Fungal/Viral | 0 [0 to 5.4] | 1.4 [0 to 7.4] | 1.5 [0 to 8.2]
  NIBSI: Bacterial/Fungal/Viral Meningitis | 0 [0 to 5.4] | 1.4 [0 to 7.4] | 0 [0 to 5.4]
  NIBSI: Respiratory Bacterial/Fungal/Viral Infection | 0 [0 to 5.4] | 0 [0 to 4.9] | 1.5 [0 to 8.2]
  CA- Major External Structural Defects | 0 [0 to 5.4] | 2.7 [0.3 to 9.5] | 0 [0 to 5.4]
  CA- Functional Defects | 0 [0 to 5.4] | 1.4 [0 to 7.4] | 0 [0 to 5.4]
  CA- Internal Structural Defects | 0 [0 to 5.4] | 1.4 [0 to 7.4] | 0 [0 to 5.4]

12. Primary Outcome: Percentage of Infant Subjects With Any SAEs
Description: SAEs assessed included any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity or is a congenital anomaly/birth defect, other situations (medical events that might jeopardize the participant or required medical/surgical intervention to prevent one of the other SAEs listed above: e.g. invasive/malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization). Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From birth to Day 43 post-birth
Population: The analysis was performed on the ESI, which included all the infants live-born to exposed maternal subjects, whose parents/LARs completed the informed consent process and signed the informed consent form.
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 22.4 [13.1 to 34.2] | 27.4 [17.6 to 39.1] | 28.8 [18.3 to 41.3]

13. Primary Outcome: Percentage of Infant Subjects With AEs Leading to Study Withdrawal
Description: as for outcome 7
Time Frame: From birth to Day 43 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

14. Primary Outcome: Percentage of Infant Subjects With Any MAEs
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Also, for instances where, due to the special circumstances, the subject could not seek medical advice for symptoms/an illness by visiting a medical facility or arranging for a home visit, the subject sought this advice instead via telephone, SMS, email, videotelephony or telemedicine, or other means. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From birth to Day 43 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 25.4 [15.5 to 37.5] | 35.6 [24.7 to 47.7] | 30.3 [19.6 to 42.9]

15. Primary Outcome: RSV MAT Immunoglobulin G (IgG)-Specific Antibody Concentrations in Terms of Geometric Mean Concentrations (GMCs) in Maternal Subjects
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by Enzyme-linked immunosorbent assay (ELISA). The corresponding antibody concentrations were expressed in ELISA units per milliliter (EU/mL) and were measured on blood samples collected from vaccinated maternal subjects.
Time Frame: At Day 1 (before vaccination), Day 31 and at delivery
Population: The analysis was performed on the Per Protocol Set-Maternal (PPSM) for immunogenicity which included all the maternal subjects who received at least 1 dose of the study intervention to which they were randomized and had post-vaccination data minus those subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 68 | 72 | 68
EU/mL
  Day 1 | 5681 [4851 to 6653] | 5837 [4962 to 6865] | 6147 [5224 to 7234]
  Day 31: number analyzed (Participants) | 58 | 68 | 60
  Day 31 | 80986 [66746 to 98263] | 105138 [93657 to 118025] | 6597 [5252 to 8288]
  Delivery: number analyzed (Participants) | 64 | 67 | 62
  Delivery | 59395 [50742 to 69524] | 59715 [51417 to 69352] | 5555 [4568 to 6755]

16. Primary Outcome: RSV-A Neutralizing Antibody Geometric Mean Titers (GMTs) in Maternal Subjects
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were expressed in Estimated Dilution 60 (ED60) and were measured on blood samples collected from vaccinated maternal subjects.
Time Frame: At Day 1 (before vaccination), Day 31 and at delivery
Population: The analysis was performed on the PPSM for immunogenicity which included all the maternal subjects who received at least 1 dose of the study intervention to which they were randomized and had post-vaccination data minus those subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 68 | 73 | 68
Titers
  Day 1 | 671.8 [544.1 to 829.4] | 694.7 [565.8 to 852.9] | 735.6 [586.7 to 922.1]
  Day 31: number analyzed (Participants) | 58 | 68 | 60
  Day 31 | 9534.2 [7758.5 to 11716.3] | 10781.2 [9150 to 12703.2] | 799.1 [622.2 to 1026.2]
  Delivery: number analyzed (Participants) | 64 | 67 | 62
  Delivery | 6162.1 [4981.2 to 7623] | 6661 [5490.7 to 8080.7] | 761.1 [612.1 to 946.3]

17. Primary Outcome: RSV MAT IgG Antibody GMCs in Infants Born to Maternal Subjects
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA. The corresponding antibody concentrations were expressed in EU/mL. The antibodies were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 3 days after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 3 days after birth
Population: The analysis was performed on the Per Protocol Set-Infants (PPSI), which included all infant subjects in the ESI who have post-delivery/birth immunogenicity data minus those who (a) were born less than 4 weeks post-maternal subject vaccination and/ or (b) have protocol deviations that lead to exclusion and for whom blood samples were collected at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 59 | 64 | 60
EU/mL | 91606.9 [76414.1 to 109820.3] | 114529.8 [100023.3 to 131140.1] | 9272.3 [7669.8 to 11209.5]

18. Primary Outcome: RSV-A Neutralizing Antibody GMTs in Infants Born to Maternal Subjects
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were presented as GMTs, expressed in ED60. The antibodies were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 3 days after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 3 days after birth
Population: The analysis was performed on the PPSI, which included all infant subjects in the ESI who have post-delivery/birth immunogenicity data minus those who (a) were born less than 4 weeks post-maternal subject vaccination and/ or (b) have protocol deviations that lead to exclusion and for whom blood samples were collected at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 60 | 64 | 61
Titers | 8414.7 [6813.4 to 10392.5] | 10262.5 [8709.9 to 12091.9] | 1244.7 [981.3 to 1578.8]

19. Primary Outcome: Geometric Mean Ratio Between Cord Blood and Maternal RSV MAT IgG-specific Antibody Concentrations
Description: The placental transfer ratio of IgG specific antibody concentration was determined from cord blood (or blood sample collected within 3 days after birth from infants if cord blood was not collected) over that of the blood sample from mother at delivery if blood sample was not collected during delivery). Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA.
Time Frame: At delivery (for maternal subjects) or within 3 days after birth (for infants)
Population: The analysis was performed on all pairs of maternal subjects (from PPSM) and their infants (from PPSI) with available results for this outcome measure at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- RSV MAT 60 Group: This group consisted of pairs of maternal subjects from RSV MAT 60- Mother Group and infant subjects from RSV MAT 60-Infants Group.
- RSV MAT 120 Group: This group consisted of pairs of maternal subjects from RSV MAT 120- Mother Group and infant subjects from RSV MAT 120-Infants Group.
- Control Group: This group consisted of pairs of maternal subjects from Control- Mother Group and infant subjects from Control-Infants Group.
Arm/Group | RSV MAT 60 Group | RSV MAT 120 Group | Control Group
Number analyzed (Participants) | 59 | 63 | 58
Ratio | 1.62 [1.44 to 1.82] | 1.9 [1.75 to 2.06] | 1.6 [1.47 to 1.75]

20. Secondary Outcome: Percentage of Maternal Subjects With Any SAE From Day 1 to Day 181 Post Delivery
Description: as for outcome 6
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 22.9 [13.7 to 34.4] | 28 [18.2 to 39.6] | 22.1 [12.9 to 33.8]

21. Secondary Outcome: Percentage of Maternal Subjects With Any MAE From Day 1 to Day 181 Post Delivery
Description: as for outcome 8
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 47.1 [35.1 to 59.4] | 53.3 [41.4 to 64.9] | 47.1 [34.8 to 59.6]

22. Secondary Outcome: Percentage of Maternal Subjects With AE Leading to Study Withdrawal From Day 1 to Day 181 Post Delivery
Description: as for outcome 7
Time Frame: From Day 1 to Day 181 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

23. Secondary Outcome: Percentage of Infant Subjects With Any SAE From Birth to Day 181 Post-birth
Description: SAEs assessed included any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject, other situations (medical events that might jeopardize the participant or required medical/surgical intervention to prevent one of the other SAEs listed above: e.g. invasive/malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization). Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 25.4 [15.5 to 37.5] | 28.8 [18.8 to 40.6] | 30.3 [19.6 to 42.9]

24. Secondary Outcome: Percentage of Infant Subjects With AE Leading to Study Withdrawal From Birth to Day 181 Post-birth
Description: as for outcome 7
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

25. Secondary Outcome: Percentage of Infant Subjects With Any MAE From Birth to Day 181 Post-birth
Description: as for outcome 8
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 40.3 [28.5 to 53] | 52.1 [40 to 63.9] | 39.4 [27.6 to 52.2]

26. Secondary Outcome: Percentage of Infant Subjects With Any SAE From Birth to Month 12 Post-birth
Description: as for outcome 23
Time Frame: From birth to Month 12 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 25.4 [15.5 to 37.5] | 28.8 [18.8 to 40.6] | 31.8 [20.9 to 44.4]

27. Secondary Outcome: Percentage of Infant Subjects With Any AE Leading to Study Withdrawal From Birth to Month 12 Post-birth
Description: An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs leading to study withdrawal = AEs identified by investigators to cause subject(s) withdrawal until the resolution of the event. These subject withdrawals were considered different from subject withdrawals for other reasons.
Time Frame: From birth to Month 12 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

28. Secondary Outcome: Percentage of Infant Subjects With Any MAE From Birth to Month 12 Post-birth
Description: as for outcome 8
Time Frame: From birth to Month 12 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 43.3 [31.2 to 56] | 57.5 [45.4 to 69] | 43.9 [31.7 to 56.7]

29. Secondary Outcome: Percentage of Maternal Subjects With RSV-associated Medically Attended Respiratory Tract Illnesses (MA-RTI)
Description: A maternal MA-RTI occurs when the maternal subject visits a healthcare professional for any respiratory symptom, including cough, sputum production and difficulty breathing. An RSV associated MA-RTI is characterised by a medically attended visit for RTI symptoms (runny nose or blocked nose or cough) and a confirmed RSV infection.
Time Frame: From delivery to Day 181 post-delivery
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of maternal subjects
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 70 | 75 | 68
Percentage of maternal subjects | 0 [0 to 5.1] | 0 [0 to 4.8] | 0 [0 to 5.3]

30. Secondary Outcome: Percentage of Infant Subjects With RSV-associated Lower Respiratory Tract Illness (LRTI)
Description: An RSV-associated LRTI is characterised by a history of cough or difficulty in breathing, a blood oxygen saturation by pulse oximetry (SpO2) lesser than (<) 95% or respiratory rate increase and a confirmed RSV infection.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 5.4] | 0 [0 to 4.9] | 0 [0 to 5.4]

31. Secondary Outcome: Percentage of Infant Subjects With RSV-associated Severe LRTI
Description: A RSV-associated severe LRTI is characterised by a history of cough or difficulty in breathing, a SpO2 < 93% or lower chest wall in-drawing and a confirmed RSV infection.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 5.4] | 0 [0 to 4.9] | 0 [0 to 5.4]

32. Secondary Outcome: Percentage of Infant Subjects With RSV-associated Very Severe LRTI
Description: A RSV-associated very severe LRTI is characterised by a history of cough or difficulty in breathing, a SpO2 < 90% or inability to feed or failure to respond/unconscious and a confirmed RSV infection.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 5.4] | 0 [0 to 4.9] | 0 [0 to 5.4]

33. Secondary Outcome: Percentage of Infant Subjects With RSV-associated Hospitalisation
Description: An RSV-associated hospitalisation is characterised by a confirmed RSV infection and a hospitalisation for an acute medical condition.
Time Frame: From birth to Day 181 post-birth
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of infant subjects
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 67 | 73 | 66
Percentage of infant subjects | 0 [0 to 5.4] | 0 [0 to 4.9] | 0 [0 to 5.4]

34. Secondary Outcome: RSV MAT IgG Antibody GMCs in Maternal Subjects, at Day 43 Post-delivery
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA. The corresponding antibody concentration were expressed in EU/mL.
Time Frame: At Day 43 post-delivery
Population: The analysis was performed on the PPSM for immunogenicity which included all the maternal subjects who received at least 1 dose of the study intervention to which they were randomized and have post-vaccination data minus those subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 53 | 59 | 50
EU/mL | 61925 [51966 to 73792] | 62871 [53878 to 73364] | 8350 [6723 to 10372]

35. Secondary Outcome: RSV-A Neutralizing Antibody GMTs in Maternal Subjects, at Day 43 Post-delivery
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were expressed in ED60.
Time Frame: At Day 43 post-delivery
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 53 | 58 | 50
Titers | 6451.3 [4842.4 to 8594.6] | 6290.7 [5000.6 to 7913.7] | 943.6 [733.4 to 1213.9]

36. Secondary Outcome: RSV-B Neutralizing Antibody GMTs in Maternal Subjects
Description: Serological assays for the determination of antibodies against RSV-B are performed by neutralization assay. The corresponding antibody titers were expressed in ED60.
Time Frame: At Day 1 (before vaccination), Day 31, at delivery and Day 43 post-delivery
Population: as for outcome 34
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother
Number analyzed (Participants) | 67 | 73 | 68
Titers
  Day 1 | 1066.3 [833.7 to 1363.9] | 1144.7 [933.1 to 1404.4] | 969.5 [790.5 to 1188.9]
  Day 31: number analyzed (Participants) | 58 | 68 | 58
  Day 31 | 13766.2 [10692.6 to 17723.2] | 15849.4 [13101 to 19174.4] | 1065.8 [846.5 to 1341.8]
  Delivery: number analyzed (Participants) | 63 | 66 | 61
  Delivery | 8983.1 [7079.7 to 11398.1] | 13335.6 [10507 to 16925.8] | 1190.7 [922.8 to 1536.5]
  Day 43 post-delivery: number analyzed (Participants) | 53 | 59 | 49
  Day 43 post-delivery | 12297.7 [9464.3 to 15979.4] | 10027.2 [8033.2 to 12516.2] | 1473.8 [1111.1 to 1954.8]

37. Secondary Outcome: RSV MAT IgG Antibody GMCs in Infants Born to Maternal Subjects, at Day 43 After Birth
Description: as for outcome 34
Time Frame: At Day 43 after birth
Population: The analysis was performed on a subcohort (subcohort V2-New borns) from PPSI, for the subjects who provided sample for this outcome measure at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 13 | 15 | 11
EU/mL | 30194.5 [18677.2 to 48813.8] | 39378.2 [33586.7 to 46168.4] | 2576.1 [1566.4 to 4236.5]

38. Secondary Outcome: RSV MAT IgG Antibody GMCs in Infants Born to Maternal Subjects, at Day 121 After Birth
Description: as for outcome 34
Time Frame: At Day 121 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 17 | 19 | 10
EU/mL | 4292.9 [3263 to 5648] | 4656.9 [3539.4 to 6127.4] | 445.5 [291.4 to 681]

39. Secondary Outcome: RSV MAT IgG Antibody GMCs in Infants Born to Maternal Subjects, at Day 181 After Birth
Description: as for outcome 34
Time Frame: At Day 181 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 11 | 19 | 11
EU/mL | 1224.1 [815.1 to 1838.4] | 1433.5 [1116.7 to 1840.1] | 179.6 [97.7 to 330.3]

40. Secondary Outcome: RSV-A Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 43 After Birth
Description: as for outcome 35
Time Frame: At Day 43 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 13 | 15 | 11
Titers | 3384.2 [2200.1 to 5205.5] | 3509.6 [2525.2 to 4877.6] | 613.3 [298.6 to 1259.8]

41. Secondary Outcome: RSV-A Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 121 After Birth
Description: as for outcome 35
Time Frame: At Day 121 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 17 | 19 | 10
Titers | 762.3 [458.3 to 1268.2] | 890.9 [648.5 to 1224] | 91.2 [56.8 to 146.5]

42. Secondary Outcome: RSV-A Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 181 After Birth
Description: as for outcome 35
Time Frame: At Day 181 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 11 | 20 | 12
Titers | 278.4 [146 to 530.9] | 324.8 [194.6 to 542.3] | 47.8 [23.8 to 96]

43. Secondary Outcome: RSV-B Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Birth
Description: Serological assays for the determination of antibodies against RSV-B were performed by neutralization assay. The corresponding antibody titers were expressed in ED60. The antibodies were measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 3 days after birth (if no cord blood sample could be obtained).
Time Frame: At delivery or within 3 days after birth
Population: The analysis was performed on the Per Protocol Set-Infants (PPSI), which included all infant subjects in the ESI who have post-delivery/birth immunogenicity data minus those who (a) were born less than 4 weeks post- maternal subject vaccination and/ or (b) have protocol deviations that lead to exclusion and for whom blood samples were collected at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 58 | 64 | 60
Titers | 13585.6 [10453.9 to 17655.4] | 18955 [15694.7 to 22892.6] | 1656.8 [1320.3 to 2079]

44. Secondary Outcome: RSV-B Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 43 After Birth
Description: Serological assays for the determination of antibodies against RSV-B were performed by neutralization assay. The corresponding antibody titers were expressed in ED60.
Time Frame: At Day 43 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 13 | 15 | 11
Titers | 5932.1 [2562.6 to 13731.7] | 6905.5 [4373.3 to 10903.8] | 548.2 [292.1 to 1028.8]

45. Secondary Outcome: RSV-B Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 121 After Birth
Description: as for outcome 44
Time Frame: At Day 121 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 17 | 19 | 10
Titers | 1119 [705.3 to 1775.4] | 1367 [950.5 to 1965.9] | 141.6 [82 to 244.6]

46. Secondary Outcome: RSV-B Neutralizing Antibody GMTs in Infants Born to Maternal Subjects, at Day 181 After Birth
Description: as for outcome 44
Time Frame: At Day 181 after birth
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
Number analyzed (Participants) | 11 | 20 | 12
Titers | 459.8 [245.9 to 859.7] | 574 [368.9 to 893.3] | 68.8 [27.1 to 174.7]

ADVERSE EVENTS:
Time Frame: For maternal groups, administration site and systemic events were collected during the 7-day follow-up period after vaccination and unsolicited adverse events during the 30-day follow-up period after vaccination. Serious adverse events were collected from Day 1 up to Month 6 post-Delivery in mothers and from Birth up to 12 months in infants.
Description: Infants born to vaccinated mothers were only monitored for AESIs and MAEs. These results are presented in the outcome measures section. Post vaccination solicited and unsolicited AEs were not collected for infants, as they were not vaccinated in the study.
Arm/Group | RSV MAT 60 Group-Mother | RSV MAT 120 Group-Mother | Control Group-Mother | RSV MAT 60 Group-Infant | RSV MAT 120 Group-Infant | Control Group-Infant
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/75 | 0/68 | 0/67 | 0/73 | 0/66
Serious Adverse Events (participants affected / at risk) | 16/70 | 21/75 | 15/68 | 17/67 | 21/73 | 21/66
Other Adverse Events (participants affected / at risk) | 56/70 | 66/75 | 47/68 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT 60 Group-Mother (N=70) | RSV MAT 120 Group-Mother (N=75) | Control Group-Mother (N=68) | RSV MAT 60 Group-Infant (N=67) | RSV MAT 120 Group-Infant (N=73) | Control Group-Infant (N=66)
Bell's palsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (4)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital acrochordon (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital arterial malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital viral hepatitis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hooded prepuce (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Naevus flammeus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Preauricular cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supernumerary nipple (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 9 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal cardiac disorder (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical cord compression (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV MAT 60 Group-Mother (N=70) | RSV MAT 120 Group-Mother (N=75) | Control Group-Mother (N=68) | RSV MAT 60 Group-Infant (N=0) | RSV MAT 120 Group-Infant (N=0) | Control Group-Infant (N=0)
Nausea (Gastrointestinal disorders) | 18 (18) | 17 (17) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 17 (18) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 13 (13) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 25 (25) | 21 (23) | 14 (14) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 40 (40) | 39 (39) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 28 (28) | 26 (28) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT04126213/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04126213/SAP_001.pdf